CLINICAL TRIAL: NCT00334243
Title: Protocol Evaluation for Improved In Vitro Fertilization Outcomes
Brief Title: Protocols for Improved in Vitro Fertilization (IVF) Outcomes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: stopped due to limited enrollment. 2 subjects were enrolled. There was NO enrollment after November 2007.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Purcell-01
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Infertility
Keywords: in vitro fertilization; infertile; infertility; pregnancy; pregnancy rates; microflare protocol; antagonist protocol; demi-halt protocol; poor responders; low antral follicle count; Infertile Patients undergoing in vitro fertilization (IVF); Patients with a previous poor response to ovarian stimulation; Patients with an antral follicle count of less than 10
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Microflare protocol for IVF
Drug: Antagonist protocol for IVF
Drug: Demi-halt protocol for IVF

SUMMARY:
Many infertile patients have a decreased chance of becoming pregnant when using in vitro fertilization (IVF). For these patients, many different treatments are available, but none of them have been shown to be better than the others. We are testing which of three different treatments are better than the others. Patients who are expected to have a decreased response to ovarian stimulation will be randomized to either a microflare protocol, an antagonist protocol, or a demi-halt protocol.

DETAILED DESCRIPTION:
Infertile patients with an anticipated poor response to ovarian stimulation will be randomized to one of three different protocols in their upcoming IVF cycle. Each of the protocols will be performed as is the standard of care with the addition of serum evaluation during the course of the stimulation as well as follicular fluid analysis which is obtained as a byproduct of the oocyte retrieval. Chart review will be performed to collect background characteristics (including age, ethnicity, previous fertility treatment), treatment response (such as oocyte number, embryo grade, embryo quality), and pregnancy outcome (such as miscarriage, singleton pregnancy, or higher-order multiple pregnancy). Statistical analysis will be performed to determine if one protocol leads to higher pregnancy rates and multivariate analysis will be performed to determine potential etiologic variables.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients
* Undergoing IVF
* Antral Follicle Count Less than 10
* Prior history of less than 5 oocytes generated during an IVF cycle

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate

SECONDARY OUTCOMES:
Cycle Cancellation Rates
Number of Oocytes Generated
Number of Embryos Generated
Serum hormonal evaluation
Follicular fluid evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle I Cedars, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States